CLINICAL TRIAL: NCT03752047
Title: Can Respiratory Rate Predict the Risk of Deterioration of Septic Patients
Status: Completed | Type: Observational
Sponsor: PMD Solutions (Industry)
Collaborators: Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: PMD-CS-006ii
Record Dates: First submitted 2018-11-20; First posted 2018-11-23 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Suspicion of Sepsis: Patients who are admitted and are diagnosed with sepsis will be recruited for this investigation.

SUMMARY:
The primary objective is to determine if the trend in Respiratory Rate measurements provided by the device under investigation can be used to predict an increase in Sequential/Sepsis-related Organ Failure Assessment (SOFA) score.

The RR trend will be measured as the difference between the RR recorded by the device at a point 15 minutes after commencement of treatment, as per the standard of care for patients suspected of being septic, and a point 3 hours following this.

DETAILED DESCRIPTION:
The primary objective is to determine if the trend in Respiratory Rate measurements provided by the device under investigation can be used to predict an increase in Sequential/Sepsis-related Organ Failure Assessment (SOFA) score.

The RR trend will be measured as the difference between the RR recorded by the device at a point 15 minutes after commencement of treatment, as per the standard of care for patients suspected of being septic, and a point 3 hours following this.

Secondary objective The secondary objective is to test if Respiratory Rate can help identify patients at increased risk of 30 day mortality.

The null Hypotheses of the planned comparison is that there is no difference in the RR trend in the 3 hours following commencement of treatment for sepsis in subjects who have an increase in SOFA score by 2 or more points and those who have a change in SOFA score of +1 or less.

The change in SOFA score will be measured at point of commencement of treatment and at 6 hours following commencement of treatment, or nearest available SOFA score determination.

Respiratory Rate captured during admission could have a predictive course for cohort of interest

The time points for reviewing the RR will be as follows:

(i) The last measurement (ii) The trend over 3 hours following commencement of treatment as per the standard of care for patients suspected of being septic.

(iii) The trend over the entire duration of admission

ELIGIBILITY:
Inclusion criteria

* ≥ 18 Years
* Admitted for a minimum of 12 hours
* Have been diagnosed with sepsis

Sepsis diagnosis confirmed by documented or suspected infection (ordering of blood culture or other microbiological investigation by the clinician) and ≥1 of the following presenting within the first 4 hours of admission:

* Fever or hypothermia, Core temperature > 38.3 or < 36 °C
* Heart rate > 90/min
* Respiratory rate > 20/min
* Altered consciousness/mental state, defined as GCS < 15
* Hyperglycemia, (BS > 6.7 mmol/L non-diabetic)
* LKC > 12 *10^9 or < 4*10^9,
* Normal LKC with > 10 % immature cells,
* CRP > highest normal local lab. Interval
* Hypotension: Systolic BP <90 mmHg, or drop in systolic BP > 40
* Hypoxemia: PaO2 < 8.5 Kpa or PaO2/FiO2 < 40 or tissue perfusion: P-lactate > 1.6
* Creatinine . 177 µmol/L
* Acute oliguria (Diuresis per hour ,0.5 ml/kg/t or 45 ml/t in 2 hours)
* Coagulopathy: Spontaneous INR > 1.5, or apt > 60 sec, thrombocytopenia
* Paralytic ileus (absence of bowel sounds)
* Hyperbilirubinemia > 34µmol/L
* Are willing to voluntarily sign a statement of informed consent to participate in this investigation

Exclusion criteria

* Allergic to medical grade skin adhesive
* Pregnant women during second and third trimester
* Continuous long term steroid use. Defined as not using steroids in the 4 weeks previous to enrolment
* Patients under the influence of substance abuse (drug or alcohol) that may interfere with their ability to cooperate and comply with the investigation procedures
* Any disorder, including cognitive dysfunction, which would affect the ability to accurately complete questionnaires and freely give full informed consent. This will be determined by the Abbreviated Mental Test Score (AMT) Cannot be followed a second time if admitted again at a later date during the study period

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: For this investigation, the population of interest are patients admitted to the Acute Medical Unit (AMU) with sepsis or that develop sepsis during their admission.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2017-03-23 (Actual); Primary Completion 2017-09-09 (Actual); Study Completion 2017-11-21 (Actual)

PRIMARY OUTCOMES:
RespiraSense triggered escalation in SOFA score | 15 minutes after commencement of treatment, as per the standard of care for patients suspected of being septic, and a point 3 hours following this.
  Escalation of SOFA score by 2 or more points. The primary endpoint will be evaluated with an ANCOVA with escalation of SOFA score by 2 or more points as a factor and mean RR in the first hour of treatment as a covariate.

SECONDARY OUTCOMES:
Upward trend in Respiratory Rate as a predictor of 30 day mortality | 30 days after discharge
  The secondary endpoint is the 30 day mortality rate after discharge.

OTHER OUTCOMES:
Upward trend in Respiratory Rate as a predictor of 30 day readmission. | 30 days after discharge
  The secondary endpoint is the 30 day readmission rate after discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of South West Jutland, Department of Emergency Medicine, Esbjerg, South West Jutland, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Data can be shared upon request.